

Prospective, Multicentric Observational Cohort Study

# **Surgical Outcomes in SPlenic Flexure CAnceRs:**

# A CompaRison of Segmental Hemicolectomy vs. Extended HemicolectOmy, and KnoWledge Assessment

**Informed Consent Form #2** 

02/12/2025

#### **Partners**



# **Volunteer Information Form**

# Surgical Outcomes in Splenic Flexure Cancer: Comparison of Segmental Hemicolectomy with Extended Hemicolectomy

#### Dear Patient,

This form has been prepared to help you make an informed decision about participating in the SPARROW Study. Please read it carefully, and do not hesitate to ask the study team any questions you may have.

#### **Background and Purpose of the Study**

Cancers of the splenic flexure represent a rare subgroup, accounting for less than 10% of all colorectal cancers. The aim of this study is to evaluate short- and long-term outcomes by comparing two different surgical approaches used for this disease (left hemicolectomy and extended right hemicolectomy). These results will be used to improve surgical decision-making and enhance patient outcomes.

## What Participation Involves

If you choose to participate in this study:

- Your treatment plan will not be altered in any way.
- Data routinely collected during your surgery and postoperative clinical care will be used.
- Participation is entirely voluntary, and you may withdraw from the study at any time without providing a reason.
- If you participate, you will be clinically monitored throughout the process.
- Total study duration: 5 years
- Expected total number of participants: 140

#### **Data to Be Collected**

- Your personal information will be anonymized and linked only to a protocol number.
- The information collected may include:
  - Age, sex, and other basic demographic data
  - Surgical details such as type of operation, duration, lymph node harvest, and any complications
  - Postoperative recovery information (e.g., time to first flatus, return to diet)



## **Risks and Benefits of Participation**

- **Risks:** There are no additional risks associated with participating in this study. All aspects of your treatment will follow current clinical standards.
- **Benefits:** Your participation may contribute to improving surgical approaches for this rare cancer type.

#### **Confidentiality and Data Security**

- All study-related data will be anonymized and stored in a way that will not reveal your identity.
- Your information will be used only by the research team and solely for the purposes of this study.
- During clinical visits, only the surgeon performing your procedure will have access to your personal medical information.

### **Your Rights**

- Participation in this study is completely voluntary.
- You have the right to refuse participation or to withdraw from the study at any time, with or without reason.
- Your decision will not affect your medical care in any way.

#### **Contact Information**

If you have any questions about the study, please feel free to contact your doctor or the research team.

#### **Consent Statement**

I have carefully read and understood the informed consent form (total of 3 pages), and my questions have been answered.

I received written and verbal explanations regarding the study mentioned above from the physician listed below.

I understand that I am volunteering to participate in this study and that I may withdraw at any time, with or without providing a reason.

I voluntarily agree to participate in this study without any pressure or coercion.



| Participant Name and Surname: Participant Signature: Date: |
|------------------------------------------------------------|
| Researcher Name and Surname: |
| Researcher Signature: |
| Date: |

